CLINICAL TRIAL: NCT02945527
Title: Open Controled Randomized Pilot Study on the Use of Acetazolamide and Dexamethasone for the Acute Phase of Perilesional Edema in Calcified Neurocysticercosis
Brief Title: Treatment of Peri-calcification Edema in Neurocysticercosis (NCC)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 62352
Record Dates: First submitted 2016-05-10; First posted 2016-10-26 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Neurocysticercosis
MeSH Terms: conditions — Neurocysticercosis | interventions — Acetazolamide; Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acetazolamide (Active Comparator): 750 mg acetazolamide p.o. divided in three dily doses, for 10 days
  Interventions: Drug: Acetazolamide
- Dexamethasone (Active Comparator): 8 mg p.o. divided in three daily daily doses, for 2 days followed by gradual tapering
  Interventions: Drug: Dexamethasone
- No additional anti-edema treatment (No Intervention): No additional treatment

INTERVENTIONS:
Drug: Acetazolamide — As described above
  Arms: Acetazolamide
Drug: Dexamethasone — As described above
  Arms: Dexamethasone

SUMMARY:
Three-arm open, randomized comparative study of acetazolamide, dexamethasone, or no additional treatment to evaluate decrease in peri-calcification edema in neurocysticercosis

DETAILED DESCRIPTION:
This study will evaluate 24 patients with calcified NCC and edema in three treatment arms to compare the reduction in edema volume

ELIGIBILITY:
Inclusion Criteria:

* Calcified NCC
* Perilesional edema on CT or MRI
* Normal lab values

Exclusion Criteria:

* Viable neurocysticercosis
* Status epilepticus
* Symptomatic intracranial hypertension
* Tuberculosis
* More than 7 days after seizure
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Decrease in Volume of Perilesional Edema Between Baseline and Day 4 | Baseline to Day 4
  MRI extension of edema

SECONDARY OUTCOMES:
Decrease in Volume of Perilesional Edema Between Baseline and Day 8 | Baseline to Day 8
  MRI extension of edema
Decrease in Volume of Perilesional Edema Between Baseline and Day 30 | Baseline to Day 30
  MRI extension of edema

CONTACTS AND LOCATIONS:
Overall Officials: Hector H. Garcia, MD, PhD, Study Chair — Universidad Peruana Cayetano Heredia
Locations (1):
- Cysticercosis Unit, Instituto Nacional de Ciencias Neurologicas, Lima, Peru

IPD SHARING:
Plan to Share IPD: No
As a concrete product, the clinical trial should provide base data to implement an affordable therapy for edema-related seizures. The data produced was going to be published in a peer reviewed journal; nevertheless, the study was prematurely terminated due to low recruitment.